CLINICAL TRIAL: NCT06017180
Title: Investigation of the Effects of Myofascial Release Techniques on Shoulder-Elbow Mobility, Sensorimotor Function and Performance in Volleyball Players
Brief Title: Effects of Myofascial Release Technique on Mobility, Sensorimotor Function and Performance in Volleyball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Fatma Özden, Physical Therapist, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 7700-GOA
Record Dates: First submitted 2022-03-21; First posted 2023-08-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Athletes; Volleyball
Keywords: foam rolling; volleyball; proprioception; upper extremity; strength; performance

STUDY DESIGN:
Intervention Model Description: intervention group and sham group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Group (Experimental): 54 healthy people playing volleyball will be included in our study and randomly divided into groups. In group I (myofascial release group), myofascial release will be applied to the shoulder and elbow region.
  Interventions: Other: Myofascial Release Techniques
- Control Group (Sham Comparator): 54 healthy people playing volleyball will be included in our study and randomly divided into groups. The sham method will be applied to the shoulder and elbow region of group II (control group).
  Interventions: Other: Sham myofascial release technique

INTERVENTIONS:
Other: Myofascial Release Techniques — Volleyball players will perform these practices with a physiotherapist 3 days a week for 8 weeks (24 sessions), and their routine sports training will continue. Participants in the group will be shown how to use rolling materials. The application will be performed as 2 sets in a session using the body weight of the person, as 10 rolls in 1 minute. The application time will be 2 minutes in total for each session. There will be 30 seconds of rest between sets. The participation rate limit for the sessions was determined as 80%. The application rate will be controlled with a metronome. The pressure to be created using body weight will be controlled by a numerical pain scale. The technique will be applied to the biceps brachii, latissimuss dorsi, upper trapezius, pectoralis minor, pectoralis major, and thoracic extensor muscles. During the application, a foam roller and a rolling stick (Thera-Band, Hygienic Corporation, Akron, OH) will be used.
  Arms: Myofascial Release Group
Other: Sham myofascial release technique — It was planned to apply the sham myofascial release technique to the athletes in the control group. In this application; with the help of the palm of the hand, pressure will be applied to the surface of the relevant muscles, first without pressure for 1 minute, then after resting for 30 seconds. The given pressure will be 2 out of 10 (0: No pain/discomfort due to pressure, 10: Unbearable pain/discomfort due to pressure). This group will also be given the right to receive a myofascial relaxation program which the experimental group received, after the study period ended.
  Arms: Control Group

SUMMARY:
Sports that require overhead activities (volleyball, tennis, basketball) include components such as rapid displacement, strength and movement control.Volleyball is also called as an overhead sport in terms of the way it is played. In the realization of these sports; Sub-parameters such as proprioceptive sense, strength, throwing rate, flexibility play a role. During these activities, the shoulder and elbow joints are overloaded. To meet this load, the joint must provide the necessary mobility and stability. Proprioceptive sense in increasing the quality and width of movement as well as providing dynamic joint stability in overhead sports; Increasing the range of motion of the joint, reducing muscle stiffness and thus increasing flexibility are effective in providing mobility. That's why it's important to develop them. Likewise, muscle strength should be increased in order to maintain movement performance and prevent injuries. The use of myofascial release techniques as an exercise method has increased in recent years. Application; The effects on parameters such as strength, performance and flexibility were investigated. Studies have focused more on the lower extremities and acute effects. There is no study on the subject examining proprioceptive sensation in volleyball players in the upper extremity. Therefore, our aim is to examine the chronic effects of the application on shoulder and elbow joint mobility, sensorimotor function and performance.

DETAILED DESCRIPTION:
Sports that require overhead activities (volleyball, tennis, basketball) include components such as rapid displacement, strength and movement control.Volleyball is also called as an overhead sport in terms of the way it is played. In the realization of these sports; Sub-parameters such as proprioceptive sense, strength, throwing rate, flexibility play a role. During these activities, the shoulder and elbow joints are overloaded. To meet this load, the joint must provide the necessary mobility and stability. Proprioceptive sense in increasing the quality and width of movement as well as providing dynamic joint stability in overhead sports; Increasing the range of motion of the joint, reducing muscle stiffness and thus increasing flexibility are effective in providing mobility. That's why it's important to develop them. Likewise, muscle strength should be increased in order to maintain movement performance and prevent injuries. Performance is the evaluation of how much the psychological, physiological and biomechanical requirements required for a sportive activity are provided. Individual and team sports, by their very nature, result in winning and losing. In this respect, it is important that the performance is at the highest level. In addition to strength, speed is also an important parameter in performance. With the programs made by combining these parameters, sportive performance and athletic success can be increased. The ability to effectively perform parameters such as throwing, throwing and hitting the ball in overhead sports affects performance results. Athletes competing in branches where overhead movements requiring high muscle activity are used intensively; In addition to strength and flexibility, which are key components of performance, sensorimotor accuracy is also of great importance.

Fascia; It is a body network that is the continuation of the connective tissue and is shaped by stretching, and it surrounds all organs and body structures. If the fascial tissue can be trained at the appropriate level (appropriate level of flexibility and elasticity), it can be beneficial in terms of protection from injuries as well as increasing sports performance. When we look at the literature, we see that the importance of this issue has increased in recent years. Myofascial release is an up-to-date method that appears to be effective in improving joint and fascia mobility, increasing body awareness, and aiding muscle reduction. Myofascial release application has become popular around the world in recent years, and it shows itself as one of the exercise trends of athletes.The use of myofascial release techniques as an exercise method has increased in recent years. Application; The effects on parameters such as strength, performance and flexibility were investigated. Studies have focused more on the lower extremities and acute effects. There is no study on the subject examining proprioceptive sensation in volleyball players in the upper extremity. Therefore, our aim is to examine the chronic effects of the application on shoulder and elbow joint mobility, sensorimotor function and performance.

With the myofascial release application that we plan to do, we aim to improve these parameters and thus provide the athletes with an alternative application method in terms of preventing injuries and improving performance. When we review the literature, we are the first study to examine the effectiveness of myofascial release in the upper extremity and the long-term effects on athletes doing overhead activities.

For all these reasons, the aim of this study is; To examine the effect of 8-week myofascial release application to the shoulder and elbow region on mobility, muscle strength, joint position sense, force matching, performance and well-being, and to examine the effect of the application at the 4th week, 8th week (end of the application), and 6th month after the first evaluation. is to detect whether there is a change in these parameters. In this study, the effect of myofascial release on shoulder and elbow joints in overhead volleyball players will be investigated for the first time. We think that our study will shed light on the studies to be done in healthy and symptomatic individuals who are interested in sports where the upper extremity is at the forefront.

ELIGIBILITY:
Inclusion criteria:

* Being playing volleyball
* Training at least two hours a week Being between the ages of 13-40
* Full active movement of the shoulder and elbow in all directions
* To have at least 3 years of overhead sports activity (volleyball) (Kurt, 2022)
* Active participation in training and competitions
* Absence of shoulder pain
* To be able to complete all the evaluations and applications to be made in the study

Exclusion criteria:

* Not wanting to participate in the study and not being able to fulfill its requirements
* History of upper extremity injury in the last 1 year
* Any history of surgery or fracture in the upper extremity
* The occurrence of pain during evaluations and applications
* Having a diagnosed disease related to the neck and shoulder
* Having any diagnosed systemic (rheumatological) musculoskeletal disease
* Have a lower extremity injury (acute and/or active) in the last six months
* Having acne and similar skin problems, open wounds that may prevent the application of rounded myofascial relaxation
* Previous application of similar rounded myofascial relaxation
* Diagnosis of diabetes mellitus and peripheral neuropathy
* Having been diagnosed with osteoporosis
* Having a diagnosis of vertigo
* Having a cardiovascular disease
* Being pregnant

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Proprioception (elbow and shoulder) | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month
  Change of biceps brachii and shoulder internal rotation joint position sense (with digital inclinometer in degree) (Target angel:Elbow:45 degree, shoulder:45 degree). The target angles to be tested will be taught by the investigators with eyes open 3 times and eyes closed 3 times. The participant will then be asked to bring it to the target angle with their eyes closed. The deviation value from the target angle will be recorded.
Muscle Strength (elbow and shoulder) | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of biceps brachii and shoulder internal rotation isometric strength (in kg, with hand held dynamometer).The average of three consecutive repetitions will be recorded.
Mobility (shoulder) | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of shoulder mobility (shoulder (internal and external rotation) range of motion, Back Scratch test:The distance between the middle fingers will be recorded in cm.). Measurements will be made 3 times, the average of the measured values will be recorded.
Performance (Speed) | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of shoulder and elbow performance (Dunk speed test with sportive radar). The tests will be conducted by measuring the maximum slam speed using a volleyball. The ball is thrown from a height of 2 to 3 meters by the coach. Participants dunk the ball into the net without touching the net and without occupying the opponent's court. Participants will be asked to practice 3 spikes at their maximum strength. The average of the three values will be taken. (km/h)

SECONDARY OUTCOMES:
Well-Being | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of participants well-being (Likert type well-being test) (Minimum:7 points, maximum: 35 points). The well-being of the participants will be evaluated with a 7-item questionnaire (fatigue, stress, sleep, muscle pain, enjoyment of training/exercise training, irritability and health). Scoring on a 5-point Likert scale will be required for each item. A total score between 7 and 35 will be calculated.
Performance | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of shoulder and elbow performance (closed kinetic chain upper extremity stability test). Participants will be in a push-up position, the distance between the two hands will be adjusted to be 90 cm, then the number of repetitions completed within 15 seconds will be recorded by extending one hand towards the other hand. The test will be repeated 3 times and the average will be taken.
Mobility | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of elbow (flexion-extension) range of motion, upper trapezius muscle length (With the test, muscle length will be recorded as short or normal) and pectoralis minor muscle length (For the pectoralis minor muscle, the length of the muscle, the distance from the junction of the sternum with the fourth rib (caudal edge) to the corocoid process, will be measured with a tape measure when the participant is standing and the upper extremity is in a free position. Three measurements will be made and the average of these measurements will be recorded in cm)
Muscle Strength | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of triceps brachii and shoulder external rotation isometric strength (in kg, with hand held dynamometer). The average of three consecutive repetitions will be recorded.
Proprioception (joint position sense and force match) | Baseline, after 4 and 8 weeks myofascial release techniques period and then follow up measurement 6. month.
  Change of shoulder external rotation and abduction joint position sense (with digital inclinometer in degree) (External rotation:45 degree, abduction:100 degree) and force match ( hand held dynamometer ) (elbow and shoulder; internal, external rotation and abduction %50 of maximum voluntary contraction) (Force match: Three maximum voluntary isometric contraction trials will be performed at the desired angles and the highest value of the three trials will be used to determine the target force. 50% of the determined value will be calculated and the participant will be asked to repeat this calculated value.) (Joint position sense: The target angles to be tested will be taught by the investigators with eyes open 3 times and eyes closed 3 times. The participants will then be asked to bring it to the target angle with their eyes closed. The deviation value from the target angle will be recorded.) The average of the three measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, PhD, Study Director — Dokuz Eylul University
Locations (2):
- Turkey (Türkiye) (2):
  - Manisa Büyük Şehir Belediyesi Spor Kulübü, Manisa
  - Manisa Gençlik ve Spor İl Müdürlüğü Voleybol Takımı, Manisa